CLINICAL TRIAL: NCT03765099
Title: Effects of Animal-Assisted Interactions (AAI) on Quality of Life in Children With Life-Threatening Conditions and Their Parents
Brief Title: Animal-Assisted Interactions in Children With Life-Threatening Conditions and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Human Animal Bond Research Institute (Unknown)
Responsible Party: Principal Investigator, Maryjo Gilmer, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC PED 18166
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Advanced Cancer; Relapsed Cancer; Refractory Cancer
MeSH Terms: conditions — Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal-Assisted Interactions (Experimental): Children and their caregivers randomly assigned to the intervention group will spend approximately 15 min with a registered canine and its owner during potentially anxiety-producing visits to the hospital.
  Interventions: Behavioral: Animal-Assisted Interactions
- Usual Care (Active Comparator): Children and their caregivers randomly assigned to the usual care group will receive usual care which may include play therapy, music therapy or visits with a social worker during their visits to the hospital.
  Interventions: Behavioral: Animal-Assisted Interactions

INTERVENTIONS:
Behavioral: Animal-Assisted Interactions — Child and caregivers randomly assigned to the intervention group will spend approximately 15 min with a registered canine and its owner during potentially anxiety-producing visits to the hospital.
  Other Names: AAI

SUMMARY:
This study will evaluate the effects of animal-assisted interactions (AAI) on stress, anxiety, and quality of life in children with a life-threatening condition and their parents. It is anticipated to be a milestone in understanding the human-animal bond.

DETAILED DESCRIPTION:
Objectives:

1. Examine the feasibility of animal-assisted interactions sessions for children with a life-threatening condition and primary caregiver to:

   * Identify and document modifications for a safe and feasible intervention,
   * Obtain recruitment estimates and determine potential recruitment barriers
   * Evaluate elements of implementation fidelity (design, training, delivery/receipt of Treatment, enactment)
   * Verify safety.

   H1-1: Children and parents (>60%) will complete the interventions and provide positive acceptability data. H1-2: Implementation fidelity can be achieved with the proposed methodology
2. Determine the preliminary efficacy of animal-assisted interactions sessions for:

   * Children with a life-threatening condition (LTC) for the outcome of health-related quality of life
   * Children with a LTC and their primary caregivers for the outcomes of stress and anxiety

H2-1 Children with a life-threatening condition who receive animal-assisted interactions will experience improved health-related quality of life (HRQOL) more than patients who do not receive animal-assisted interactions.

H2-2a Children with life-threatening condition who receive animal-assisted interactions will experience decreased stress and anxiety more than parents of children who do not receive animal-assisted interactions.

H2-2b Primary caregivers of children with a life-threatening condition who receive animal-assisted interactions will experience decreased stress and anxiety more than parents of children who do not receive animal-assisted interactions.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-17 years old
* Confirmed diagnosis of relapsed or refractory cancer

Exclusion Criteria:

* Reported fear or anxiety of dogs (child or parent)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life | up to 3 months
  The Peds Quality of Life measure will be administered to children and their parents (proxy) once a month
Anxiety | up to 3 months
  The state-trait anxiety inventory will be administered to children and their parents after each intervention or usual care visit
Stress | up to 3 months
  Saliva samples to measure cortisol levels will be administered to children after animal-assisted interventions or after completion of measures in usual care group

CONTACTS AND LOCATIONS:
Overall Officials: Maryjo Gilmer, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mahoney AB, Akard TF, Cowfer BA, Dietrich MS, Newton JL, Gilmer MJ. Impact of Animal-Assisted Interaction on Anxiety in Children With Advanced Cancer and Their Caregivers. J Palliat Med. 2024 Jan;27(1):75-82. doi: 10.1089/jpm.2023.0091. Epub 2023 Sep 25. PMID 37751186
- [Derived] Cowfer BA, Akard TF, Gilmer MJ. Animal-Assisted Interventions for Children with Advanced Cancer: Child and Parent Perceptions. Palliat Med Rep. 2021 Nov 17;2(1):328-334. doi: 10.1089/pmr.2021.0039. eCollection 2021. PMID 34927159

DOCUMENTS (1):
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03765099/ICF_000.pdf